CLINICAL TRIAL: NCT02223143
Title: A Registration Study for Primary and Secondary Prevention in Dyslipidemic Taiwanese
Brief Title: A Registration Study for Dyslipidemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200910021R
Record Dates: First submitted 2014-08-18; First posted 2014-08-22 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Atherosclerotic Vascular Diseases
Keywords: Lipid lowering therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Cardiovascular disease (CVD), including coronary heart disease (CHD) and stroke, is a leading cause of morbidity and mortality. Dyslipidemia has long been recognized to be the most important risk factor in the development of atherosclerosis in human beings. In Taiwan, the rates for hypercholesterolemia (≧250mg/dl) were 4.3% and 5.5% in 1970; 12.99% in 1980; and 17.1% in 1990. Those for hypertriglyceridemia (≧200 mg/dl) were 6.5% and 11.1% in 1970 and 13.0% in 1990. Low serum HDL-C was an isolated and independent coronary risk factor among a good number of Taiwanese people. Lowering of low-density lipoprotein cholesterol (LDL-C) with statins has in the last decade become part of the standard treatment regimen in patients with dyslipidemia. However, most embarrassing, is the insufficient data for clinical use in Taiwan. It is necessary to have rationalized and balanced guideline for the management of dyslipidemia in Taiwan, based on our local epidemiological, clinical and basic research data. Because all these trials were conducted in Caucasians and no large-scaled end-point research about the lipid lowering therapy (LLT) was published in Asians before, this registry study attempts to define the status of lipid lowering therapy in Taiwan and the effect of LLT on CVD morbidity and mortality in a large population of patients receiving primary or secondary prevention therapy. The medications will only depend on the decision made by the primary care physicians. The patient or physician can decide to be withdrawn from this registry at any time because of any reason. The lipid profile change, myopathy, or liver enzyme change after the LLT will also be recorded.

DETAILED DESCRIPTION:
This is a registry study to define the status of lipid lowering therapy in Taiwan and the effect of LLT on CVD morbidity and mortality in a large population of patients receiving primary or secondary prevention therapy. The medications will only depend on the decision made by the primary care physicians. The patient or physician can decide to be withdrawn from this registry at any time because of any reason.

All potential patients will be screened for the eligibility in a screening visit. Those who fill the inclusion criteria at screening will be invited for the registry study into different groups. The follow-up will take place yearly thereafter for 5 years, through clinical visiting, phone follow-up, or records from the NHIB Taiwan. At each clinical visit, vital signs, clinical endpoints, adverse events, concurrent medication information and laboratory specimens will be obtained as complete as possible. With phone or records from NHIB, only clinical endpoints will be recorded. If the primary care physician intends to treat the patient's lipid profile to the target, he/she can add, delete or adjust the LLT by his/her clinical judgement.

ELIGIBILITY:
Inclusion Criteria:

* One with atherosclerotic vascular diseases
* One without ASVD but with at least 1 CV risk factor
* Apparent healthy persons

Exclusion Criteria:

* One with hemodynamically significant valvular or congenital heart disease
* One with any non-cardiovascular diseases which may affect prognosis

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All potential patients will be screened for the eligibility in a screening visit. Those who fill the inclusion criteria at screening will be invited for the registry study into different groups.
Sampling Method: Probability Sample
Enrollment: 35000 (Estimated)
Dates: Start 2009-01; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
The time to first occurrence of a major cardiovascular event | up to 5 years
  The major CV (cardiovascular) event will be defined as CV death, hospitalization for nonfatal MI (myocardial infarction) or stroke, or cardiac arrest with resuscitation

SECONDARY OUTCOMES:
Composite cardiovascular outcome | up to 5 years
  The composite cardiovascular (CV) outcome will be any CV events (any major CV events plus hospitalization for any revascularization procedure, unstable angina, or congestive heart failure, and peripheral arterial disease, defined as new clinical diagnosis or hospitalization for such disease). In addition, individual components of the composite end points will be also prespecified as secondary outcomes, as will all-cause mortality.

OTHER OUTCOMES:
The biochemistry change | up to 5 years
  The tertiary objective of this trial is to evaluate the biochemistry change of lipid profile change, myopathy, or liver enzyme change after the lipid lowering therapy.

CONTACTS AND LOCATIONS:
Overall Officials: C C W, Principal Investigator — chauchungwu@ntu.edu.tw
Locations (1):
- NTUH, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes